CLINICAL TRIAL: NCT00003800
Title: Correlation of Histopathology, Immunohistochemistry and Quantitative Radiology With Outcome in Early Stage Nonseminomatous Germ Cell Tumor
Brief Title: Diagnostic Study of Patients With Stage I Testicular Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000066944; U10CA021115 (NIH); ECOG-8897
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Testicular Germ Cell Tumor
Keywords: stage I malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor; testicular yolk sac tumor and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Carcinoma, Embryonal | interventions — Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laboratory/CT evaluation (No Intervention): Observation following orchiectomy
  Interventions: Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: radionuclide imaging

INTERVENTIONS:
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: radionuclide imaging

SUMMARY:
RATIONALE: Diagnostic procedures may improve a doctor's ability to predict the recurrence of testicular cancer.

PURPOSE: Diagnostic trial to detect the risk of recurrent disease in patients who have stage I testicular cancer and who have undergone orchiectomy within the previous 12 weeks.

DETAILED DESCRIPTION:
OBJECTIVES:

* Use histopathological and immunohistological analysis of the primary testis tumor along with quantitative radiographic assessment to identify a subset of patients with clinical stage I nonseminomatous germ cell tumor of the testis who have a very low risk of metastasis.
* Compare these findings with other predictive models of risk of metastasis after orchiectomy in this group of patients.

OUTLINE: Patients undergo primary retroperitoneal lymph node dissection (RPLND) or active surveillance as management of their disease. The choice of treatment is determined by the physician and the patient. Patients with pathologically positive resected lymph nodes may undergo treatment (observation or adjuvant chemotherapy) at investigator's discretion.

All patients are tested by quantitative radiology and blood markers (HCG and AFP) at baseline and then at various times after surgery to identify pathologic stage II disease. The timing of these studies depends on the stage of disease and/or type of disease management.

Patients who undergo RPLND, have stage I or II disease, and do not receive adjuvant therapy (radiation or chemotherapy) are followed monthly during year 1, every 2 months during year 2, every 6 months during years 3-5, and annually thereafter.

Patients who undergo RPLND, have stage II disease, and receive adjuvant therapy are followed every 2 months during year 1, every 4 months during year 2, every 6 months during years 3-5, and annually thereafter.

Patients who do not undergo RPLND are followed monthly during year 1, every other month during year 2, every 6 months during years 3-5, and annually thereafter.

PROJECTED ACCRUAL: A total of 315 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinical stage I nonseminomatous germ cell tumor of the testis
* Must have had a radical inguinal orchiectomy with or without retroperitoneal lymph node dissection within prior 12 weeks

  * AFP and HCG normal or decreasing after orchiectomy at a rate consistent with known half lives
  * Pathology blocks and radiologic studies available
* No metastatic disease on physical exam or chest or abdominal/pelvic CT
* No pure seminoma (unless associated with elevated AFP at diagnosis)

PATIENT CHARACTERISTICS:

Age:

* 15 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No prior malignancy including prior primary testicular cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Ages: 15 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 1999-11-16 (Actual); Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Evidence of regional or metastatic spread | observed at least annually
  Patients with putative stage A non-seminomatous germ cell tumors are assessed at baseline using chest xray and blood markers. They are then followed monthly during year 1, every 2 months during year 2, twice a year during years 3-5, and annually thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Foster, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (12):
- United States (12):
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - Scott and White Hospital, Temple, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin